CLINICAL TRIAL: NCT05544084
Title: Adaptation and Implementation of a Patient Navigation Program for Cervical Cancer Screening Across Contexts in Senegal
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Illinois at Chicago (Other)
Responsible Party: Principal Investigator, Jon Andrew Dykens, Associate Professor of Family and Community Medicine, University of Illinois at Chicago
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Screening
Other Study IDs: R01CA258683 (NIH)
Record Dates: First submitted 2022-09-12; First posted 2022-09-16 (Actual); Last update posted 2025-03-13 (Actual); Status verified 2025-03

CONDITIONS: Cervical Cancer; Behavior
MeSH Terms: conditions — Uterine Cervical Neoplasms; Behavior

STUDY DESIGN:
Intervention Model Description: Conduct an effectiveness-implementation hybrid type 1 stepped-wedge randomized pragmatic trial of the adapted patient navigation program across Kedougou and Dakar, Senegal.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Adapted Patient Navigation Program (Experimental): Adaptation of a patient navigation approach to effect change in cervical cancer screening uptake in Kedougou and Dakar, Senegal. Conduct a stepped-wedge randomized pragmatic trial in three districts in the Kedougou Region and three districts in Dakar to evaluate the impact of The Adapted Program. In order to conduct this trial, investigators will deploy The Adapted Program and evaluate the impact of The Adapted Program on screening uptake and time to treatment initiation (for those with abnormal screening results) within the various contexts across clusters. Investigators will also explore the effect of The Adapted Program on intrapersonal- and community-level barriers. Finally, evaluate the implementation outcomes of The Adapted Program within the context of these rural and urban districts, whereby clusters serve as their own controls as they cross over from the control to intervention group.
  Interventions: Behavioral: Patient Navigator Approach
- Control (No Intervention): Standard of care

INTERVENTIONS:
Behavioral: Patient Navigator Approach — Patient navigators in collaboration with community health workers will work with women eligible for cervical cancer screening to overcome intrapersonal and community level barriers to screening in order to engage early with the health system for cervical cancer screening and follow-up of positive screens. Their support can help patients get the cancer screenings and follow-up care they need, while addressing prevalent gender inequities and community-level stigma associated with cancer within the Senegal context.
  Arms: Adapted Patient Navigation Program

SUMMARY:
The goal of this project is to prevent unnecessary deaths due to cervical cancer in Senegal. This mixed methods research responds to identified intrapersonal- and community-level barriers to early cervical cancer screening uptake, follow-up, and treatment among women there. Investigators will apply the Dynamic Adaptation Process (DAP) as integrated into the Exploration, Preparation, Implementation, Sustainment (EPIS) framework to study the adaptation of an evidence-based cervical cancer patient navigation program in urban and rural contexts in Senegal, measure the intervention effectiveness, and evaluate programmatic implementation outcomes. By studying the process of adaptation of a patient navigation program in a low- and middle-income country (LMIC), investigators will build new knowledge while addressing an important public health issue. The project demonstrates innovation by advancing both adaptation and implementation process knowledge of an evidence-based patient navigation intervention in various contexts within a LMIC with a particular focus on how the adaptation responds to cancer-related stigma, misinformation, and women's autonomy in healthcare decision-making. Investigators will build knowledge through local learning which will further the long-term goal to inform the national cervical cancer prevention and control programs in two areas of Senegal and other similar LMICs.

DETAILED DESCRIPTION:
The goal of this project is to prevent unnecessary deaths due to cervical cancer in Senegal. This mixed methods research responds to identified intrapersonal- and community-level barriers to early cervical cancer screening uptake, follow-up, and treatment among women in Senegal. Investigators will apply the Dynamic Adaptation Process to study the adaptation of an evidence-based cervical cancer patient navigation program in urban and rural contexts of Senegal, measure the intervention effectiveness, and evaluate programmatic implementation outcomes.

Aim 1: Evaluate the adaptation process of the evidence-based Chinatown Patient Navigation Program utilizing the Dynamic Adaptation Process across rural and urban contexts in Kedougou and Dakar, Senegal. (n=6 clusters)

Aim 2: Conduct an effectiveness-implementation hybrid type 1 stepped-wedge randomized pragmatic trial of the adapted patient navigation program across Kedougou and Dakar, Senegal.

H1 - Participants who receive active navigation services will be more likely to get screened for cervical cancer (primary outcome) and obtain treatment more rapidly. (n=370 women) H2 - Participants who receive patient navigation services and their partners will experience or report fewer intrapersonal- and community-level barriers including cancer-related stigma (secondary outcomes) and lack of autonomy in healthcare decision-making. (n=740 women and men)

Aim 3: Evaluate the implementation outcomes9 (feasibility, acceptability, fidelity, penetrance, sustainability, and cost) of The Adapted Patient Navigation Program across multiple contexts in the Kedougou and Dakar regions, using mixed methods and guided by the Exploration, Preparation, Implementation, Sustainment (EPIS) Framework.(n=96 participants across 6 clusters)

Aim 1 will adapt the evidence-based Chicago Chinatown Program into the urban and rural Senegal contexts. Investigators will accomplish the EXPLORATION PHASE of Aim 1 by first conducting a multilevel (system/ organization, provider, and client) assessment of stakeholder characteristics relevant to the context of three districts in rural Kedougou and three districts in urban Dakar, Senegal (randomly selected). Contextual assessment will be iterative, capturing data at each interval of the stepped wedge approach. This will continue to inform the iterative adaptation of the program. In the PREPARATION PHASE, investigators will delineate the core elements and adaptable features of the Chinatown Program and describe the iterative adaptation (guided and ad hoc), through a participatory approach, of The Adapted Program across Kedougou and Dakar, Senegal. Next, in the IMPLEMENTATION PHASE, Aim 2, investigators will conduct a stepped-wedge randomized pragmatic trial in three districts in the Kedougou Region and three districts in Dakar to evaluate the impact of The Adapted Program. In order to conduct this trial, investigators will deploy The Adapted Program and evaluate the impact of The Adapted Program on screening uptake and time to treatment initiation (for those with abnormal screening results) within the various contexts across clusters. Investigators will also explore the effect of The Adapted Program on intrapersonal- and community-level barriers. Finally, during the SUSTAINMENT PHASE Aim 3 investigators will evaluate the implementation outcomes of The Adapted Program within the context of these rural and urban districts. Investigators will evaluate the feasibility, acceptability, fidelity, penetrance, sustainability, and cost of The Adapted Program as each district prepares, rolls out, and sustains The Adapted Program in the Kedougou and Dakar regions.

Each of the six clusters completes all four Implementation steps (exploration, preparation, implementation, and sustainment), with extensive initial support from research team members during exploration, preparation, and implementation. Support decreases gradually as clusters gain the experience to sustain patient navigation activities. If successful, the health system will integrate patient navigation as a means to facilitate the uptake of cervical cancer services and manage patients along the cancer care continuum. Evaluation of the success of patient navigation is determined as follows:

For Aims 1 and 3, the Exploration, Preparation, Implementation, Sustainment (EPIS) framework guides the mixed methods analysis of success and contextual factors related to success.

For Aim 2, investigators assess outcomes four times using participants' self-report surveys and medical records.

At a time of major global health policy shifts, these results will provide strong evidence for patient navigation policy decisions in low-income countries and will advance implementation science.

ELIGIBILITY:
Inclusion Criteria:

The inclusion criteria for samples a, b, & c are as follows:

1) Senegal citizen between the ages of 25 and 69, 2) willing to participate in survey assessments;

The additional criteria apply for both women and men for the follow samples:

Sample a: 3) an invited member of the study National Advisory Board or Regional Implementation Resource Teams as defined above; 4) able to read and write in French.

Sample b: 3) employed by the state at a study site health facility as a patient navigator, clinician (nurse, midwife) who treats and educates patients, or is a community health worker at the facility or community level (Bajenu Gox - women's health educator).

Sample c: Women: 3) a woman living with a male partner who also agrees to participate in the study, 4) eligible to seek cervical cancer prevention services at a designated health facility in Senegal. Men: 3) a man living in a household with at least one woman eligible to seek cervical cancer prevention services at a designated health facility in Senegal.

Exclusion Criteria:

* No additional exclusion criteria exist.

Ages: 25 Years to 69 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — No exclusions will be made on the basis of gender for the baseline or longitudinal individual surveys or focus groups. However, focus groups will be split by gender indication (e.g., women-only focus group)
Enrollment: 901 (Estimated)
Dates: Start 2023-08-01 (Actual); Primary Completion 2026-05-01 (Estimated); Study Completion 2027-05-01 (Estimated)

PRIMARY OUTCOMES:
Change in the number of women screened for the first time, age stratified uptake through self-report questionnaire and confirmed through record review | Baseline and then every 12 months through 36 months
  Change in the number of women reporting cervical cancer screening uptake, age stratified

SECONDARY OUTCOMES:
Change in time to treatment for dysplasia, age stratified, through record review | Baseline and then every 12 months through 36 months
  Change in the time from diagnosis of a positive cervical cancer screen to treatment for dysplasia, age stratified
Change in perceived stigma of cervical cancer as the fault of the individual, through questionnaire | Baseline and then every 12 months through 36 months
  Change in the number of women and men stating that if a woman gets cervical cancer it is probably their own fault, age stratified
Change in decision to get cervical cancer screen, age stratified, through questionnaire | Baseline and then every 12 months through 36 months
  Change in the number of women and men stating that women are able to make their own decisions regarding getting screened for cervical cancer, age stratified
Change in awareness of cervical cancer, age stratified, through questionnaire | Baseline and then every 12 months through 36 months
  Change in the number of women and men stating awareness of cervical cancer, age stratified"
Change in knowledge of need for screen despite symptoms, age stratified, through questionnaire | Baseline and then every 12 months through 36 months
  Change in the number of women and men stating awareness of the necessity for cervical cancer screening despite having no symptoms, age stratified
Change in spouse communication about cervical cancer screening, through questionnaire | Baseline and then every 12 months through 36 months
  Perception of men and women of open communication with spouse regarding healthy approach to cervical cancer screening for women.

CONTACTS AND LOCATIONS:
Overall Officials: Jon A Dykens, MD, MPH, Principal Investigator — University of Illinois at Chicago
Locations (1):
- University of Cheikh Anta Diop, Institute of Health and Development, Dakar, Senegal

IPD SHARING:
Plan to Share IPD: Yes
Investigators will share all IPD that underlie results in a publication
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: Upon completion of the study. The materials will be available indefinitely.

REFERENCES:
- [Background] Ongtengco N, Thiam H, Collins Z, De Jesus EL, Peterson CE, Wang T, Hendrix E, Ndiaye Y, Gueye B, Gassama O, Kasse AA, Faye A, Smith JS, Fitzgibbon M, Dykens JA. Role of gender in perspectives of discrimination, stigma, and attitudes relative to cervical cancer in rural Senegal. PLoS One. 2020 Apr 28;15(4):e0232291. doi: 10.1371/journal.pone.0232291. eCollection 2020. PMID 32343755
- [Background] Dykens JA, Linn AM, Irwin T, Peters KE, Pyra M, Traore F, Toure Diarra M, Hasnain M, Wallner K, Linn P, Ndiaye Y. Implementing visual cervical cancer screening in Senegal: a cross-sectional study of risk factors and prevalence highlighting service utilization barriers. Int J Womens Health. 2017 Jan 27;9:59-67. doi: 10.2147/IJWH.S115454. eCollection 2017. PMID 28184171
- [Background] Simon MA, Tom LS, Leung I, Wong E, Knightly EE, Vicencio DP, Yau A, Ortigara K, Dong X. The Chinatown Patient Navigation Program: Adaptation and Implementation of Breast and Cervical Cancer Patient Navigation in Chicago's Chinatown. Health Serv Insights. 2019 Apr 18;12:1178632919841376. doi: 10.1177/1178632919841376. eCollection 2019. PMID 31037032